CLINICAL TRIAL: NCT05162105
Title: Quick Returns - Sleep, Cognitive Functions and Individual Differences: An Experimental Approach
Brief Title: Quick Returns - Sleep, Cognitive Functions and Individual Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 303671
Record Dates: First submitted 2021-08-30; First posted 2021-12-17 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Shift Work Schedule; Sleep Deprivation
Keywords: Shift Work; Quick Return; Sleep; Cognitive Performance; Circadian Rhythm; Genotype; Shift Work Tolerance
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to the QR-condition (evening shift followed by a day shift) or a day shift followed by another day shift. After a four week wash-out, participants return to work in the opposite condition.
Who Masked: Participant
Masking Description: Participants will not be provided information regarding hypotheses or expected results from the different conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evening shift followed by day shift (Quick Return) (Experimental): Participants work a simulated evening shift, from 03:00PM to 11:00PM, followed by a simulated day shift, 07:00AM to 03:00PM, the following day.
  Interventions: Other: Short rest (8 hour) between two consecutive shifts.
- Day shift followed by day shift (Active Comparator): Participants work a simulated day shift, from 07:00AM to 03:00PM, followed by another simulated day shift, from 07:00AM to 03:00PM, the following day.
  Interventions: Other: 16 hour rest opportunity between to consecutive shifts.

INTERVENTIONS:
Other: Short rest (8 hour) between two consecutive shifts. — Participants will have shortened rest opportunity (8 hours) between two consecutive shifts, due to the shift work schedule.
  Arms: Evening shift followed by day shift (Quick Return)
Other: 16 hour rest opportunity between to consecutive shifts. — Participants will have a 16 hour rest opportunity between shifts, due to shift work schedule.
  Arms: Day shift followed by day shift

SUMMARY:
The project will contribute with new knowledge concerning how short rest periods between two consecutive shifts (<11h, often defined as a Quick Return (QR)) affects sleep and cognitive performance. The study will further examine whether individual differences in personality traits and genotypes may explain individual differences in performance and sleep. Data will be collected with a randomized cross-over design, in an experimental laboratory setting.

DETAILED DESCRIPTION:
Rotating shift workers may have a narrow time window to rest after an evening shift, before returning early to work for a day shift. In the literature, a rest opportunity of less than 11 hours between two consecutive shifts, is defined as a Quick Return (QR). Most often, this is occurs when working an evening shift followed by a day shift. Survey- and longitudinal studies have found associations between QRs and an increased risk of being involved in occupational accidents. However, no studies have experimentally investigated how a QR scenario may affect performance at work and sleep between the two shifts. Thus, the project will experimentally simulate QRs, where a battery of cognitive tests will be administered in a laboratory to indicate performance. Objective and subjective sleep will be measured/reported at home where participants normally sleep. Additionally, genotype- and personality trait data will be collected and used as moderators in the analyses.

A randomized cross-over design with two groups will be applied. In one condition, participants will work an evening shift (03:00PM-11:00PM) followed by a day shift (07:00AM-03:00PM, QR). In the other condition, participants work a day shift (07:00AM-03:00PM) followed by another day shift. Four weeks later after being in one of the conditions, the participants will return to the laboratory and work in the opposite condition. Sleep will be subjectively reported with a sleep diary and objectively measured using a low-powered ultra-wideband radar, two days before and between the two simulated shifts in each of the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants are physically and mentally healthy (assessed with BMI and 'General Health Questionnaire-12)'.
* Participants accept to comply to the protocol (retain regular bed- and wake times before the simulated shifts).
* Refrain from alcohol and maintain regular nicotine and caffeine usage during participation.
* Norwegian as primary language/proficiency in Norwegian language.

Exclusion Criteria:

* Neurological, psychiatric or sleep related disorders ('Bergen Insomnia Scale, 'Global sleep assessment questionnaire').
* Extreme 'morning-eveningness' type ('Horne-Östberg).
* Use of medication that affect sleep or cognitive performance.
* Pregnancy.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Sustained Attention | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Sustained attention will be measured using the Psychomotor Vigilance Test (PVT). The PVT is a commonly used test to assess the effect of sleep deprivation on cognitive functioning. The test will be conducted every 1.5h - 2h during simulated shifts, in total five times during the day shift (07:30AM, 09:00AM,10:30AM, 12:30PM and 02:30PM) and five times during the evening shift (03:30PM, 05:00PM, 6:30PM, 8:30PM and 10:30PM).
Sleepiness | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  The Karolinska Sleepiness Scale (KSS) is a single item question measuring sleepiness on a likert scale from 1 - 9 ('1' - "Extremely alert" to '9' - "Very sleepy/fighting sleep"). The test will be conducted every 1.5h - 2h during simulated shifts, in total five times during the day shift (07:30AM, 09:00AM,10:30AM, 12:30PM and 02:30PM) and five times during the evening shift (03:30PM, 05:00PM, 6:30PM, 8:30PM and 10:30PM).
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Sleep Onset Latency' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'sleep onset latency' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Sleep Onset Latency in the two sleep opportunities will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Total Sleep Time' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'total sleep time' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy). Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Total Sleep Time in the two sleep opportunities will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Time in Light Sleep' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'time in light sleep' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Time in Light Sleep in the two sleep opportunities will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Time in Deep Sleep' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'time in deep sleep' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Time in Deep Sleep in the two sleep opportunities will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Time in Rapid Eye Movement(REM)-sleep' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'time in REM-sleep' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Time in Rapid Eye Movement(REM)-sleep in the two sleep opportunities will be compared.

SECONDARY OUTCOMES:
Mood/Affect | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Mood/affect is measured using the Positive and Negative Affect Scale (PANAS). PANAS contains 20 items. Each item is rated on a likert scale from 1 to 5 ('1' - None" and '5' - Extremely"). The test will be conducted every 1.5h - 2h during simulated shifts, in total five times during the day shift (07:30AM, 09:00AM,10:30AM, 12:30PM and 02:30PM) and five times during the evening shift (03:30PM, 05:00PM, 6:30PM, 8:30PM and 10:30PM).
Moral Decision | Difference between day 2, in simulated QR (evening- followed by day shift) and day 2 in the control condition (day- followed by day shift). Day 2 in QR- and control combination: 7AM-3PM.
  The Defining Issue Test (DIT-2) will be used to evaluate the effect of simulated short rest between two shifts (QR) on morality (decision making). DIT-2 presents five moral dilemmas where participants rate and rank issues surrounding the dilemmas on a likert scale from 1 to 5 ('1' - "Very important" to '5' - "Very little important"). Will be completed once at the start of each shift.
Change in Cognitive Throughput | Changes from first to last test session on day 2 in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2 in the control condition (day- followed by day shift). Day 2 in QR- and control combination: 7AM-3PM.
  Cognitive throughput will be measured using the 'digit symbol substitution task'. Taken throughout the shifts every 1.5h - 2h in total 5 times during each day shift (07:30AM, 09:00AM,10:30AM, 12:30PM and 02:30PM) and five times during the evening shift (03:30PM, 05:00PM, 6:30PM, 8:30PM and 10:30PM).
Selective Attention | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Selective attention will be measured using a 'visual search task'. The test will be taken twice per simulated shift; once during first half and once during second half of the shift.
Executive functioning | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Executive functioning will be measured using the 'attentional network task'. The test will be taken twice per simulated shift; once during first half and once during second half of the shift.
Dexterity | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Dexterity will be measured using the 'grooved pegboard test'. The test will be taken twice per simulated shift; once during first half and once during second half of the shift.
Verbal Memory | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Verbal memory will be measured using a 'word probe recall test'. The test will be taken twice per simulated shift; once during first half and once during second half of the shift.
Cognitive Inhibition | Changes from first to last test session on day 2, in a simulated QR (evening- followed by day shift) and changes from first to last test session on day 2, in the control condition (day- followed by day shift). Day 2 both combinations: 7AM-3PM.
  Cognitive inhibition will be measured using the 'go/no-go' test. The test will be taken twice per simulated shift; once during first half and once during second half of the shift.
Individual Differences - Mini International Personality Item Pool (Mini-IPIP) | Pre-intervention
  To examine if individual differences can moderate a potential effect of short rest between two shifts, Mini IPIP will be used. Mini-IPIP is a 20-item short form of the 50-item International Personality Item Pool-Five Factor Model. Scores participant on five dimensions: neuroticism, extraversion, agreeableness, conscientiousness, and openness based on a set of likert-scale questions from 1 - 5 ('1' - "Very incorrect" to '5' - "Very correct").
Individual Differences - Dark Triad Personality Scale | Pre-intervention
  To examine if individual differences can moderate a potential effect of short rest between two shifts, the Dark Triad Personality scale will be used. Dark Triad Personality Scale contains 12-items. The test scores the participant based on a set of likert-scale questions from 1 - 9 ('1'- "Completely disagree" to '9' "Completely agree") on the dimensions; machiavellianism, narcissism and psychopathy.
Individual Differences - Revised Circadian Type Inventory (CTI-R) | Pre-intervention
  To examine if individual differences can moderate a potential effect of short rest between two shifts, the CTI-R will be used. CTI-R contains 11-items indicating ability to change sleeping rhythm based on the dimensions; flexibility and languidity. The test scores the participant on based on a set of likert-scale questions from 1 - 5 ('1' - "Almost never" to '5' - "Almost always"). High scores on flexibility reflect better ability to sleep and work at odd times, whereas high scores on languidity indicates difficulties overcoming drowsiness and feeling of lethargy following sleep loss.
Individual Differences - Horne-Östberg Morning-Eveningness Questionnaire (MEQ) | Pre-intervention
  To examine if individual differences can moderate a potential effect of short rest between two shifts, the MEQ will be used. MEQ contains 19-items indicating circadian preference; morning-/evening type.
Individual Differences - Genotypes | Pre-intervention
  To examine if individual differences can moderate a potential effect of short rest between two shifts, saliva samples will be collected to analyze for genotypes related to shift work tolerance.
  Genotyping will be done with regard to: SLC6A4 tandem repeat length in the promoter (short; S versus long; L), rs25531 (A versus G), rs8192440, rs12506228 and rs4680. Analyses will be done using Custom TaqMan genotyping assays.
Arousal prior to bedtime - one night between two day shifts versus one night between evening- followed by day shift | Prior to bedtime the night between the two shifts in the QR condition (from 11PM-7AM) compared to the night between two shifts in the control condition (from 3PM-7AM).
  Pre-Sleep Arousal Scale (PSAS) will be used to examine if participants differ in arousal-level at bedtime in the two sleep opportunities. PSAS contains 16 items, each being rated on a 5-point likert scale from 1 to 5 ('1' - "Not at all" to '5' - "Extremely"). Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Arousal at bedtime in the two sleep opportunities in each condition will between will be compared.
Subjective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Sleep Quality' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'sleep quality' is reported in a sleep diary. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Sleep quality in the two sleep opportunities will be compared.
Subjective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Wake After Sleep Onset' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'wake after sleep onset' is reported in a sleep diary. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Wake after sleep onset in the two sleep opportunities will be compared.
Subjective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Sleep Efficiency' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'sleep efficiency' is reported in a sleep diary. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Sleep efficiency in the two sleep opportunities will be compared.
Subjective Sleep,one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Sleep Onset Latency' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'sleep onset latency' is reported in a sleep diary. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Sleep Onset Latency in the two sleep opportunities will be compared.
Subjective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Bedtime' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'bedtime' is reported in a sleep diary. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Bedtime in the two sleep opportunities between will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Wake after sleep onset' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'wake after sleep onset' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Wake after sleep onset in the two sleep opportunities will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Sleep Efficiency' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'sleep efficiency' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Sleep Efficiency in the two sleep opportunities will be compared.
Objective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Bedtime' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'bedtime' will be objectively measured using a low-powered ultra -wideband Xethru sleep radar (Somnofy), placed next to the bed. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Bedtime in the two sleep opportunities will be compared.
Subjective Sleep, one sleep opportunity between day- followed by day shift versus one sleep opportunity between evening- followed by day shift - 'Total Sleep Time' | Sleep taking place between the two days in the QR condition (from 11PM-7AM) compared to sleep taking place between the two days in the control condition (from 3PM-7AM).
  To evaluate the effect of simulated short rest between two shifts (QR) on sleep, 'total sleep time' is reported in a sleep diary. Sleep opportunity will in the QR-condition be between 11PM-7AM and in the control-condition between 3PM-7AM, as a consequence of simulated shift schedule (QR-condition; first shift on day 1 occurring 3PM-11PM & second shift on day 2 occurring 7AM-3PM. Control-condition; first shift on day 1 occurring 7AM-3PM & second shift on day 2 occurring 7AM-3PM the following day). Total sleep time in the two sleep opportunities will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Department of Psychosocial Science, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
After the project has ended the data will be anonymized and no direct recognizable information will be stored.

REFERENCES:
- [Derived] Holmelid O, Harris A, Pallesen S, Bjorvatn B, Vedaa O, Waage S, Nielsen MB, Djupedal ILR, Sunde E. Acute effects of a simulated quick return on subjective sleepiness, mood, and cognitive performance: A laboratory crossover controlled trial. Chronobiol Int. 2024 Aug;41(8):1116-1127. doi: 10.1080/07420528.2024.2380736. Epub 2024 Jul 22. PMID 39037118